CLINICAL TRIAL: NCT01871441
Title: A Two Step Approach to Haploidentical Hematopoietic Stem Cell Transplantation for Patients in Remission From HLA Partially-Matched Related Donors-Effect of Maternal Donors on Outcomes
Brief Title: Haploidentical Donor Hematopoietic Stem Cell Transplant in Treating Patients With Hematologic Malignancies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial was closed due to poor accrual.
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13D.127; 2012-104 (Other: CCRRC); JT 3048 (Other: JeffTrial Number)
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Results first posted 2018-01-09 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Whole-Body Irradiation; Cyclophosphamide; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (haploidentical allogeneic HSCT) (Experimental): Patients undergo TBI BID on days -9 to -6, undergo DLI on day -6, and receive cyclophosphamide IV over 2 hours on days -3 and -2.
  TRANSPLANT: Patients undergo haploidentical allogeneic hematopoietic stem cell transplant on day 0.
  GVHD PROPHYLAXIS: Patients receive tacrolimus IV beginning on day -1 with taper beginning on day 42, and mycophenolate mofetil IV BID from day -1 to day 28.
  Interventions: Radiation: Total-body irradiation; Biological: Donor lymphocytes infusion (DLI); Drug: Cyclophosphamide; Procedure: Allogeneic hematopoietic stem cell transplantation (HSCT); Drug: Tacrolimus; Drug: Mycophenolate mofetil

INTERVENTIONS:
Radiation: Total-body irradiation — Undergo TBI
  Other Names: TBI
Biological: Donor lymphocytes infusion (DLI) — Undergo DLI
  Other Names: Allogeneic Lymphocytes; ALLOLYMPH
Drug: Cyclophosphamide — Given IV
  Other Names: Endoxan; Cytoxan; Neosar; Procytox; Revimmune; cytophosphane
Procedure: Allogeneic hematopoietic stem cell transplantation (HSCT) — Undergo haploidentical allogeneic HSCT
Drug: Tacrolimus — Given IV
  Other Names: FK-506; fujimycin; Prograf; Advagraf; Protopic
Drug: Mycophenolate mofetil — Given IV
  Other Names: CellCept; Myfortic; MMF

SUMMARY:
This phase II trial studies how well haploidentical donor hematopoietic stem cell transplant works in treating patients with hematologic malignancies. Giving chemotherapy and total-body irradiation before a donor stem cell transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. Giving an infusion of the donor's T cells (donor lymphocyte infusion) may replace the patient's immune cells and help destroy any remaining cancer cells. When the stem cells from a related donor, that closely matches the patient's blood, are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Examine the 1 year disease free survival (DFS) rate of patients with maternal donors or sibling donors who share the maternal haplotype (maternal group) and compare them to patients receiving cells from donors who have points from other characteristics such as killer immunoglobulin-like receptor (KIR) ligand mismatching, minor histocompatibility antigen (MHag) differences, or number of human leukocyte antigen (HLA) mismatches (non-maternal group).

SECONDARY OBJECTIVES:

I. Assess the incidences of relapse and graft-versus-host disease (GVHD) in maternal recipients whose only eligible donors are offspring.

II. Assess the incidence of grades III-IV GVHD in female recipients with male donors.

III. Compare the rates of DFS in recipient-donor combinations in which there is at least 1 KIR ligand mismatch versus those without a KIR ligand mismatch.

OUTLINE:

Patients undergo total body irradiation (TBI) twice daily (BID) on days -9 to -6, undergo donor lymphocyte infusion (DLI) on day -6, and receive cyclophosphamide intravenously (IV) over 2 hours on days -3 and -2.

TRANSPLANT: Patients undergo haploidentical allogeneic hematopoietic stem cell transplant on day 0.

GVHD PROPHYLAXIS: Patients receive tacrolimus IV beginning on day -1 with taper beginning on day 42, and mycophenolate mofetil IV BID from day -1 to day 28.

After completion of study treatment, patients are followed up at 90, 180, and 270 days, and 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient with a hematologic or oncologic diagnosis without morphological evidence of disease in which allogeneic HSCT is thought to be beneficial.
2. Patients must have a related donor who is a two or more allele mismatch at the HLA-A; B; C; DR loci.
3. Patients must have adequate organ function:

   1. LVEF (Left ventricular ejection fraction) of >50%
   2. Diffusion Capacity for Carbon Monoxide (DLCO) >50% of predicted corrected for hemoglobin
   3. Adequate liver function as defined by a serum bilirubin <1.8, Aspartate Aminotransferase (AST) or alanine aminotransferase (ALT) < 2.5X upper limit of normal
   4. Creatinine clearance of > 60 ml/min
4. Performance status > 80% (TJU Karnofsky)
5. Hematopoietic Comorbidity Index (HCT-CI) Score < 5 Points
6. Patients must be willing to use contraception if they have childbearing potential
7. Able to give informed consent, or if decisionally impaired, have a legal next of kin or guardian that can give informed consent

Exclusion Criteria:

1. Performance status < 80 % (TJU Karnofsky)
2. HCT-CI Score > 5 Points
3. Combination of Performance status of < 80% (TJU Karnofsky) and an HCT-CI of 4 points or more.
4. HIV positive
5. Active involvement of the central nervous system with malignancy
6. Psychiatric disorder that would preclude patients from signing an informed consent
7. Pregnancy
8. Patients with life expectancy of < 6 months for reasons other than their underlying hematologic/oncologic disorder
9. Patients who have received alemtuzumab within 8 weeks of the transplant admission, or who have recently received horse or rabbit anti-thymocyte globulin and have an ATG level of > 2 ugm/ml
10. Patients who cannot receive cyclophosphamide
11. Patients with evidence of another malignancy, exclusive of a skin cancer that requires only local treatment, should not be enrolled on this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-05-17 (Actual); Primary Completion 2013-12-12 (Actual); Study Completion 2016-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dolores Grosso, DNP, CRNP, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Haploidentical Allogeneic HSCT): Patients undergo TBI BID on days -9 to -6, undergo DLI on day -6, and receive cyclophosphamide IV over 2 hours on days -3 and -2.
  TRANSPLANT: Patients undergo haploidentical allogeneic hematopoietic stem cell transplant on day 0.
  GVHD PROPHYLAXIS: Patients receive tacrolimus IV beginning on day -1 with taper beginning on day 42, and mycophenolate mofetil IV BID from day -1 to day 28.
  Total-body irradiation: Undergo TBI
  Donor lymphocytes infusion (DLI): Undergo DLI
  Cyclophosphamide: Given IV
  Allogeneic hematopoietic stem cell transplantation (HSCT): Undergo haploidentical allogeneic HSCT
  Tacrolimus: Given IV
  Mycophenolate mofetil: Given IV
Period: Overall Study
Arm/Group | Treatment (Haploidentical Allogeneic HSCT)
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Haploidentical Allogeneic HSCT)
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (11.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Disease-free Survival (DFS)
Description: Disease free survival (DFS), defined as the time to death, relapse or disease progression.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Haploidentical Allogeneic HSCT)
Number analyzed (Participants) | 4
Participants | 1

2. Secondary Outcome: Number of Participants With Relapse of Disease
Description: Relapse of Disease is defined as the return of a disease or the signs and symptoms of a disease after a period of improvement. Relapse is almost always associated with the immunological failure of the donor immune system to recognize and/or respond to reemergence of a tumor. The number of participants with relapse of disease will be collected.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Haploidentical Allogeneic HSCT)
Number analyzed (Participants) | 4
Participants | 2

3. Secondary Outcome: Rate of Grade III-IV GVHD in Female Recipients With Male Donors
Description: The rates of grade III-IV GVHD in female recipients with male donors will be computed with corresponding exact binomial 95% confidence intervals.
Time Frame: Up to 1 year
Population: No data were collected or analyzed.
Arm/Group | Treatment (Haploidentical Allogeneic HSCT)
Number analyzed (Participants) | 0

4. Secondary Outcome: The Rates of Grade III-IV GVHD in Female Recipients With Male Donors Will be Computed With Corresponding Exact Binomial 95% Confidence Intervals.
Description: The difference in DFS in recipient-donor combinations in which there is at least 1 KIR ligand mismatch versus those without a KIR ligand mismatch will be tested using log-rank test.
Time Frame: Up to 1 year
Population: No data were collected or analyzed.
Arm/Group | Treatment (Haploidentical Allogeneic HSCT)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Treatment (Haploidentical Allogeneic HSCT)
All-Cause Mortality (participants affected / at risk) | 3/4
Serious Adverse Events (participants affected / at risk) | 4/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Haploidentical Allogeneic HSCT) (N=4)
increased LFTs (Hepatobiliary disorders) | 1 (1)
Colitis - infectious diarrhea (Gastrointestinal disorders) | 1 (1)
Fever (Immune system disorders) | 2 (2)
CMV reactivation (Immune system disorders) | 1 (1)
UTI (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Haploidentical Allogeneic HSCT) (N=4)
Abdominal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Acid reflux (Gastrointestinal disorders) | 1 (1)
Anxiety (Nervous system disorders) | 3 (3)
Arrhythmia (Cardiac disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Awakening to Urinate (General disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Blurred vision (Eye disorders) | 2 (2)
C. Difficile (Infections and infestations) | 1 (1)
CMV reactivation (Immune system disorders) | 1 (1)
Constipation (Reproductive system and breast disorders) | 3 (3)
Dehydration (General disorders) | 2 (2)
Depression (Nervous system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (5)
Dizziness (General disorders) | 1 (1)
Dry Hands (Skin and subcutaneous tissue disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (2)
Dysgeusia (General disorders) | 1 (1)
Electrolyte Abnormalities (General disorders) | 2 (2)
Elevated transaminase (Blood and lymphatic system disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Fever (Infections and infestations) | 4 (8)
Fluid overload (General disorders) | 2 (2)
GERD (Gastrointestinal disorders) | 1 (1)
Glaucoma (Eye disorders) | 1 (1)
Hallucinations (Nervous system disorders) | 1 (1)
Hives - related to injection (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Cardiac disorders) | 3 (3)
Hypotension (Cardiac disorders) | 2 (3)
Increased Creatinine (Blood and lymphatic system disorders) | 1 (2)
Increased LFTs (Renal and urinary disorders) | 2 (2)
Indigestion (Gastrointestinal disorders) | 1 (1)
Insomnia (Nervous system disorders) | 1 (1)
Iron overload (Blood and lymphatic system disorders) | 1 (1)
Itching (Skin and subcutaneous tissue disorders) | 1 (1)
Knee pain (General disorders) | 1 (1)
Swelling (General disorders) | 1 (1)
Lightheadedness (General disorders) | 1 (1)
Mucositis (General disorders) | 3 (3)
Numbness (Nervous system disorders) | 1 (1)
Parotiditis (General disorders) | 1 (1)
Pericatheter Thrombus (Renal and urinary disorders) | 1 (1)
Pruitis (Skin and subcutaneous tissue disorders) | 2 (5)
Pronatriuretic Peptide elevated (General disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rigors (Musculoskeletal and connective tissue disorders) | 1 (1)
Runny nose (General disorders) | 1 (1)
Short term memory loss (Nervous system disorders) | 1 (1)
Sweating (General disorders) | 1 (1)
Swollen hands (General disorders) | 1 (1)
SOB (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stomach cramping (Gastrointestinal disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (3)
Tachypenea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Trouble sleeping (General disorders) | 2 (3)
Twitching (Nervous system disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Watery Eyes (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes